CLINICAL TRIAL: NCT01675401
Title: Vascular Function Markers: Differences Between Lean and Abdominally Overweight / Obese Men and Effects of Weight Loss
Brief Title: Body Weight and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MEC 12-3-040
Record Dates: First submitted 2012-08-21; First posted 2012-08-30 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Body Weight; Obesity; Weight Loss; Vascular Function Markers
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Body Weight; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight-loss treatment (Experimental): A very-low energy diet (Modifast Intensive) for 4-5 weeks providing 2.1 MJ/day in order to reduce body weight. After 4-5 weeks a mixed solid energy-restricted diet up to 4.2 MJ/day with a recommended composition for the following 1-2 weeks. Then, a diet matching their energy requirements to maintain newly achieved body weights (weight-stable conditions) for at least 2 weeks.
  Interventions: Other: Weight-loss treatment
- No-weight loss treatment (Other): Maintenance of habitual diet and physical activity for 8 weeks to maintain body weights.
  Interventions: Other: No-weight loss treatment

INTERVENTIONS:
Other: Weight-loss treatment — A very-low energy diet (Modifast Intensive) for 4-5 weeks providing 2.1 MJ/day in order to reduce body weight. After 4-5 weeks a mixed solid energy-restricted diet up to 4.2 MJ/day with a recommended composition for the following 1-2 weeks. Then, a diet matching their energy requirements to maintain newly achieved body weights (weight-stable conditions) for at least 2 weeks.
  Arms: Weight-loss treatment
Other: No-weight loss treatment — Maintenance of habitual diet and physical activity for 8 weeks to maintain body weights.
  Arms: No-weight loss treatment

SUMMARY:
An increased body mass impairs vascular function (VF), an important characteristic of subjects suffering from type 2 diabetes and a risk marker for cardiovascular diseases. However, a wide variety of in vivo VF markers exists each measuring different aspects of VF. Each of these markers addresses a different aspect of the vasculature. Studies comparing under standardized conditions the differences and relationships of the many different VF measurements in lean and abdominally overweight / obese subjects are missing. Also, there is a great need to know which of these markers are sensitive to dietary challenges.

Therefore, it is imperative to conduct an extensive study on dietary effects and interrelationships of a broad spectrum of VF measurements and plasma biomarkers in lean and overweight / obese subjects. Focus will be on FMD, a well accepted biomarker for cardiovascular disease. The investigators propose to examine, in a two-way parallel-randomized human intervention study, the effects of weight-loss in abdominally overweight / obese men on VF markers and plasma biomarkers related to low-grade inflammation and vascular activity during the fasting and both the postprandial and hyperinsulinemic state. Furthermore, differences - and relations between - VF measurements and plasma biomarkers will be compared cross-sectionally between lean and abdominally overweight / obese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Waist circumference below 94 cm (lean subjects) or between 102 - 110 cm (abdominally overweight / obese subjects)
* Caucasian
* Plasma glucose < 7.0 mmol/L
* Serum total cholesterol < 8.0 mmol/L
* Serum triacylglycerol < 4.5 mmol/L
* Plasma HbA1c < 6.5%
* No current smoker
* No diabetic patients
* No familial hypercholesterolemia
* No abuse of drugs
* Less than 14 alcoholic consumptions per week
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* No use of medication known to affect blood pressure, serum lipid or glucose metabolism
* No severe medical conditions that might interfere with the study, such as epilepsy, asthma, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* No active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* No contra-indications for MRI imaging
* Willingness to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Women
* Non-caucasian
* Plasma glucose ≥ 7.0 mmol/L
* Serum total cholesterol ≥ 8.0 mmol/L
* Serum triacylglycerol ≥ 4.5 mmol/L
* Plasma HbA1c ≥ 6.5%
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 14 alcoholic consumptions per week
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Use of use of medication known to affect blood pressure, serum lipid or glucose metabolism
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Contra-indications for MRI imaging
* Use of an investigational product within the previous 1-month
* Not willing to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study, during the study or for 4 weeks after completion of the study
* Not or difficult to venipuncture as evidenced during the screening visit

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Vascular activity: differences between lean and abdominally overweight / obese men and effects of weight loss | Difference after weight-loss due to restriction of energy intake for 8 weeks and change from baseline at 2 hours after meal consumption
  Flow-mediated dilation (FMD) of the brachial artery.

SECONDARY OUTCOMES:
Vascular function markers related to the macrovasculature: differences between lean and abdominally overweight / obese men and effects of weight loss | Difference after weight-loss due to restriction of energy intake for 8 weeks and change from baseline during the postprandial (at 2 hours after meal consumption) / hyperinsulinemic state (at 2 hours after initiation of the clamp)
  Carotid-wall intima-media thickness (IMT), carotid compliance and distensibility, pulse wave velocity and analysis (PWV and PWA) and peripheral artery tonometry (PAT).
Vascular function markers related to the microvasculature: differences between lean and abdominally overweight / obese men and effects of weight loss | Difference after weight-loss due to restriction of energy intake for 8 weeks and change from baseline during the postprandial (at 1 and 3 hours after meal consumption) / hyperinsulinemic state (at 2 hours after initiation of the clamp)
  Capillary video microscopy of the finger skin, skin microvascular vasomotion, glycocalyx thickness, retina photography, skin auto fluorescence and contrast enhanced ultrasound (CEUS) in skeletal muscle.
Metabolic risk markers related to the metabolic syndrome: differences between lean and abdominally overweight / obese men and effects of weight loss | Difference after weight-loss due to restriction of energy intake for 8 weeks and change from baseline during the postprandial (during 4 hours after meal consumption) / hyperinsulinemic state (during 3 hours after initiation of the clamp)
  Biomarkers for low-grade inflammation and endothelial activation.

OTHER OUTCOMES:
Body fat components and fat content of intra-abdominal organs: differences between lean and abdominally overweight / obese men and effects of weight loss | Difference after weight-loss due to restriction of energy intake for 8 weeks
  Dixon MRI measurements in order to quantify abdominal fat compartments (i.e. subcutaneous and visceral fat) and fat content of abdominal organs (i.e. liver).
Blood pressure: difference between lean and abdominally overweight / obese men and effects of weight loss | Difference after weight-loss due to restriction of energy intake for 8 weeks
  24-hr ambulatory blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Mensink, PhD, Principal Investigator — Maastricht University Medical Center; Casper G Schalkwijk, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Van den Eynde MDG, Kusters YHAM, Houben AJHM, Scheijen JLJM, van Duynhoven J, Fazelzadeh P, Joris PJ, Plat J, Mensink RP, Hanssen NMJ, Stehouwer CDA, Schalkwijk CG. Diet-induced weight loss reduces postprandial dicarbonyl stress in abdominally obese men: Secondary analysis of a randomized controlled trial. Clin Nutr. 2021 May;40(5):2654-2662. doi: 10.1016/j.clnu.2021.03.042. Epub 2021 Apr 15. PMID 33933731
- [Derived] Joris PJ, Plat J, Kusters YHAM, Houben AJHM, Stehouwer CDA, Schalkwijk CG, Mensink RP. Effects of diet-induced weight loss on postprandial vascular function after consumption of a mixed meal: Results of a randomized controlled trial with abdominally obese men. Clin Nutr. 2020 Oct;39(10):2998-3004. doi: 10.1016/j.clnu.2020.01.006. Epub 2020 Jan 13. PMID 31982191
- [Derived] Fazelzadeh P, Hoefsloot HCJ, Hankemeier T, Most J, Kersten S, Blaak EE, Boekschoten M, van Duynhoven J. Global testing of shifts in metabolic phenotype. Metabolomics. 2018 Oct 4;14(10):139. doi: 10.1007/s11306-018-1435-8. PMID 30830386
- [Derived] Telgenkamp I, Kusters YHAM, Schalkwijk CG, Houben AJHM, Kooi ME, Lindeboom L, Bons JAP, Schaper NC, Joris PJ, Plat J, Mensink RP, Stehouwer CDA, Brouwers MCGJ. Contribution of Liver Fat to Weight Loss-Induced Changes in Serum Hepatokines: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2719-2727. doi: 10.1210/jc.2018-02378. PMID 30753672
- [Derived] Schutten MTJ, Kusters YHAM, Houben AJHM, Scheijen JLJM, van de Waarenburg MPH, Schalkwijk CG, Joris PJ, Plat J, Mensink RP, de Leeuw PW, Stehouwer CDA. Aldosterone Is Not Associated With Metabolic and Microvascular Insulin Sensitivity in Abdominally Obese Men. J Clin Endocrinol Metab. 2018 Feb 1;103(2):759-767. doi: 10.1210/jc.2017-01541. PMID 29211893
- [Derived] Kusters YH, Schalkwijk CG, Houben AJ, Kooi ME, Lindeboom L, Op 't Roodt J, Joris PJ, Plat J, Mensink RP, Barrett EJ, Stehouwer CD. Independent tissue contributors to obesity-associated insulin resistance. JCI Insight. 2017 Jul 6;2(13):e89695. doi: 10.1172/jci.insight.89695. eCollection 2017 Jul 6. PMID 28679946
- [Derived] Joris PJ, Plat J, Kusters YH, Houben AJ, Stehouwer CD, Schalkwijk CG, Mensink RP. Diet-induced weight loss improves not only cardiometabolic risk markers but also markers of vascular function: a randomized controlled trial in abdominally obese men. Am J Clin Nutr. 2017 Jan;105(1):23-31. doi: 10.3945/ajcn.116.143552. Epub 2016 Nov 23. PMID 27881395